CLINICAL TRIAL: NCT00826215
Title: A Randomized Controlled Trial of the Long-Term Efficacy of Electroacupuncture for Chronic Neck Pain
Brief Title: Electroacupuncture for Chronic Neck Pain
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hong Kong Baptist University (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Dr. Shi Ping Zhang, School of Chinese Medicine, Hong Kong Baptist Universtiy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04060191
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: Neck Pain
Keywords: mechanical; neck pain; chronic; acupuncture; chronic mechanical neck pain
MeSH Terms: conditions — Neck Pain; Bronchiolitis Obliterans Syndrome | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Electroacupuncture treatment
  Interventions: Device: electroacupuncture
- 2 (Sham Comparator): Sham laser acupuncture
  Interventions: Device: Sham laser acupuncture

INTERVENTIONS:
Device: electroacupuncture — Nine sections of 45 minutes electroacupuncture treatment in three weeks
  Arms: 1
Device: Sham laser acupuncture — Sham laser acupuncture
  Arms: 2

SUMMARY:
Objective: The primary objective of this study is to evaluate the long-term efficacy of electroacupuncture for chronic neck pain. The secondary objective is to document any possible side effects of acupuncture.

Design and Subjects: Prospective, randomised controlled trial comparing the outcomes of treatment and placebo interventions. Subjects are 200 adult patients with chronic mechanical neck pain.

Setting: Outpatient clinics.

Interventions: Patients will be randomly allocated to one of the two groups receiving either: electroacupuncture (real treatment) or placebo (sham laser acupuncture). Each treatment will last for 45 minutes. Each patient will receive a total of nine treatments (three times per week for three weeks).

Main outcome measures:

Primary outcome measures: Neck pain disability index (Northwick Park Neck Pain Questionnaire).

Secondary outcome measures: Maximum pain related to motion on visual analogue scale. Quality of life (SF-36). Use of medication. Sick leave because of neck pain. Treatment-related adverse effects, such as pain, skin irritation, bleeding and dizziness, will also be assessed.

Assessments will be made before treatment, one month, three months and six months after the treatment course. The credibility of placebo treatment will also be assessed.

Expected results: We expect that patients in the treatment group will have significant improvements on primary and secondary outcome measures, when compared with patients in the inert placebo group.

Conclusion: This study will provide credible evidence regarding whether electroacupuncture is effective in reducing chronic neck pain. Patients, healthcare professionals, and government policy makers can make use of this information to improve clinical outcomes and reduce costs

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female subjects age above 18 with mechanical neck pain for over three months.

Exclusion Criteria:

* Patients who have received acupuncture treatment for any purpose in the last 6 months.
* Patients who will be unlikely to attend all treatment sessions.
* Patients with systemic diseases, such as diabetes or cardiovascular disorder.
* Patients with a history of traumatic injury of the neck or upper back from T1-T6, precious fracture or surgery to the neck, neurological deficits (e.g., muscle weakness or changes in spinal reflex jerks), a history of malignancy, congenital abnormality of the spine, or systemic bone and joint disorders (e.g., RA).
* Patients who are seeking compensation for neck-related condition.
* Patients who have needle phobia.
* Pregnant and breast feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-02 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Change in neck pain specific disability index as measured by the Northwick Park Neck Pain Questionnaire (NPQ). | 6 months

SECONDARY OUTCOMES:
i) Change in maximum pain related to motion, regardless the direction of movement. ii) Quality of life as assessed by SF-36 health survey. iii) Use of medication because of neck pain iv) Sick leave because of neck pain. | 6 months
Adverse effects. | 6 months